CLINICAL TRIAL: NCT02634060
Title: Home basEd faecaL calProtectin Measurements Predicting Adalimumab Induction Destiny
Acronym: HELP-AID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Belgian Inflammatory Bowel Disease Research and Development (BIRD) VZW (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: S58392
Record Dates: First submitted 2015-12-14; First posted 2015-12-17 (Estimated); Last update posted 2024-06-27 (Actual); Status verified 2017-10

CONDITIONS: Crohn Disease; Colitis, Ulcerative
Keywords: adalimumab; fecal calprotectin; home based
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Home Based Fecal Calprotectin (Experimental): IBDoc® at week 0, 4 and 8 using smartphone. All material will be provided by the third party The same stool sample of the home base faecal calprotectin will be brought to the hospital and used for ELISA faecal calprotectin measurement at week 0, 4 and 8 for UC patients and week 0 and 4 for CD patients.
  IBDoc® results will be forwarded to the patient and the health care professional.
  Interventions: Device: Home Based Fecal Calprotectin

INTERVENTIONS:
Device: Home Based Fecal Calprotectin — Home Based Fecal Calprotectin measurement at weeks 0, 4 and 8
  Other Names: IBDoc

SUMMARY:
Recently a smartphone application IBDoc® was developed to enable patients to measure faecal calprotectin at home in an easy way. In this HELP-AID trial we want to evaluate the value of these home based IBDoc® faecal calprotectin measurements in predicting short- and mid-term outcome to ADA induction therapy in patients with moderate-to-severe IBD.

Patients known with moderate-to-severe CD and ulcerative colitis starting ADA therapy will be asked to participate in this study. They will be asked to collect a stool sample at 3 different time points (week 0, 4 and 8). This faecal sample needs to be loaded on a test cassette with an extraction device. In a second step, the patient can turn his smartphone into an easy to use test cassette reader by taking a picture and using the CalApp® which is based on an immunochromatographic test. Finally, the CalApp® will transmit the test results securely to the health care professional.

In this study we want to evaluate the predictive value of absolute and relative faecal calprotectin values measured by IBDoc® on clinical, biological and endoscopic outcome at week 12. Furthermore, we want to evaluate the correlation between IBDoc® and classical ELISA measurements of faecal calprotectin, and the convenience of this system to the patient and the health care professional.

DETAILED DESCRIPTION:
Adalimumab (Humira®), a fully human monoclonal antibody to TNF, has been given an important position in the treatment of patients with an inflammatory bowel disease (IBD). However, not all patients respond adequately to this relatively expensive and potentially toxic therapy. Adapting the standard treatment regimen to the individual needs of the patient may favor the short and long term outcome of this therapy.

Following daily clinical practice, patients will receive standard induction therapy with 160 mg adalimumab at week 0, followed by 80 mg adalimumab at week 2. Starting at week 4 patients will receive a maintenance therapy with 40 mg adalimumab every other week. If a patient shows an insufficient response, the dose can be increased to 40 mg adalimumab every week.

Defining predictors of response to ADA has become a major objective in scientific research. One of the predictors of response may be an early decrease in faecal calprotectin. Faecal calprotectin is a protein which presence in the stool of a patient correlates with endoscopic disease activity. A persistently elevated faecal calprotectin after start up with adalimumab treatment may suggest that this patient needs a higher dose.

Recently a smartphone application IBDoc® was developed to enable patients to measure faecal calprotectin at home in an easy way. In this HELP-AID trial we want to evaluate the value of these home based IBDoc® faecal calprotectin measurements in predicting short- and mid-term outcome to ADA induction therapy in patients with moderate-to-severe IBD.

Patients known with moderate-to-severe CD and ulcerative colitis starting ADA therapy will be asked to participate in this study. They will be asked to collect a stool sample at 3 different time points (week 0, 4 and 8). This faecal sample needs to be loaded on a test cassette with an extraction device. In a second step, the patient can turn his smartphone into an easy to use test cassette reader by taking a picture and using the CalApp® which is based on an immunochromatographic test. Finally, the CalApp® will transmit the test results securely to the health care professional.

In this study we want to evaluate the predictive value of absolute and relative faecal calprotectin values measured by IBDoc® on clinical, biological and endoscopic outcome at week 12. Furthermore, we want to evaluate the correlation between IBDoc® and classical ELISA measurements of faecal calprotectin, and the convenience of this system to the patient and the health care professional.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age;
* Established diagnosis of UC or CD for at least 3 months, with histopathological confirmation available in the record of the patient;
* Patients having failed steroids or immunomodulatory therapy for at least 3 months, or being intolerant to this therapy;
* Patients should have moderate-to-severe disease at baseline, defined as For CD: an Harvey-Bradshaw-Index above 7 and a C-reactive protein of at least 5 mg/L; For UC: a total Mayo score of at least 6 and an endoscopic sub-score of at least 2;
* Latent tuberculosis excluded within 3 months prior to ADA therapy using Chest X-ray and IFNγ release assay or tuberculin skin test; or adequate treatment for latent tuberculosis initiated for at least four weeks in case of positive screening;
* The patients should have a smartphone and be able to use a new smartphone application;
* Written informed consent must be obtained and documented;

Exclusion Criteria:

* Diagnosis of IBD type unclassified (IBDU);
* Previous (procto)colectomy for UC;
* Patients with an ostomy;
* Previous therapy with ADA;
* Patients with CD with a baseline CRP < 5mg/L at baseline;
* Patients with CD and absence of luminal disease;
* Patient with UC lacking faecal blood loss (Mayo bleeding score 0);
* Patients with UC with an ileal pouch-anal or ileo-rectal anastomosis
* Patients with acute severe IV steroid refractory colitis;
* Patients with any condition that would prevent completion of the study including history of drug or alcohol abuse, history of mental illness, or history of noncompliance with treatments or visits;
* Patients with absolute or relative contraindications for anti-TNF therapy, including intra-abdominal collections, symptomatic strictures, demyelinating disease, heart failure, …;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2016-03-31; Primary Completion 2018-06-01 (Actual); Study Completion 2022-09-05 (Actual)

PRIMARY OUTCOMES:
In UC: Steroid-free mucosal healing (Mayo 0 or 1) at week 8 without prior need for ADA dose optimization, taking into account all kind of topical and systemic steroids. | Week 8
  The predictive value of an early faecal calprotectin amelioration (EFCA) measured by IBDoc between baseline and week 4, in predicting steroid-free mucosal healing (Mayo 0 or 1) at week 8 without prior need for ADA dose optimization, taking into account all kind of topical and systemic steroids. EFCA is defined as a decrease in faecal calprotectin measured by IBDoc between baseline and week 4 with at least 80% or a faecal calprotectin less than 50 μg/g at week 4.
In CD: Steroid-free clinical remission at week 12, defined as an Harvey-Bradshaw-Index <5 and a C-reactive protein <5 mg/L, without prior need for ADA dose optimization and taking into account all kind of topical and systemic steroids | Week 12
  The predictive value of EFCA measured by IBDoc® between baseline and week 4, in predicting steroid-free clinical remission at week 12 , defined as an Harvey-Bradshaw-Index <5 and a C-reactive protein <5 mg/L, without prior need for ADA dose optimization and taking into account all kind of topical and systemic steroids. EFCA is defined as a decrease in faecal calprotectin measured by IBDoc® between baseline and week 4 with at least 80% or a faecal calprotectin less than 50 μg/g at week 4.

SECONDARY OUTCOMES:
In UC: The predictive value of an absolute and relative faecal calprotectin measured by IBDoc® between baseline and week 4 | 4 weeks
  The predictive value of an absolute and relative faecal calprotectin measured by IBDoc® between baseline and week 4 in predicting:
  * steroid-free complete mucosal healing (Mayo 0) at week 8, and week 26, without prior need for ADA dose optimization;
  * steroid-free mucosal healing (Mayo 0 or 1) at week 26, without prior need for ADA dose optimization;
  * steroid-free clinical response (decrease from baseline in the total Mayo score ≥3 and ≥30% with a decrease in the rectal bleeding sub-score of ≥1 point or an absolute rectal bleeding sub-score 0 or 1) at week 8, week 12, and week 26, without prior need for ADA dose optimization;
  * steroid-free clinical remission (Mayo ≤2, no individual sub-score >1) at week 8, week 12, and week 26, without prior need for ADA dose optimization;
  * ADA treatment optimization;
  * ADA treatment discontinuation;
In UC: The predictive value of an absolute and relative faecal calprotectin measured by IBDoc® between baseline and week 8 | 8 weeks
  The predictive value of an absolute and relative faecal calprotectin measured by IBDoc® between baseline and week 8 in predicting:
  * steroid-free complete mucosal healing (Mayo 0) at week 26, without prior need for ADA dose optimization;
  * steroid-free mucosal healing (Mayo 0 or 1) at week 26, without prior need for ADA dose optimization;
  * steroid-free clinical response (decrease from baseline in the total Mayo score ≥3 and ≥30% with a decrease in the rectal bleeding sub-score of ≥1 point or an absolute rectal bleeding sub-score 0 or 1) at week 12, and week 26, without prior need for ADA dose optimization;
  * steroid-free clinical remission (Mayo ≤2, no individual sub-score >1) at week 12, and week 26, without prior need for ADA dose optimization;
  * ADA treatment optimization;
  * ADA treatment discontinuation;
In CD: The predictive value of an absolute and relative faecal calprotectin measured by IBDoc® between baseline and week 4 | 4 weeks
  The predictive value of an absolute and relative faecal calprotectin measured by IBDoc® between baseline and week 4 in predicting:
  * steroid-free clinical-remission at week 26, without prior need for ADA dose optimization;
  * steroid-free clinical response (HBI <5 or drop in HBI with ≥3) at week 12, and week 26, without prior need for ADA dose optimization;
  * steroid-free biological remission (CRP <5 mg/L) at week 12, and week 26, without prior need for ADA dose optimization;
  * steroid-free biological response (CRP <5 mg/L or drop with ≥50%) at week 12, and week 26;
  * ADA treatment optimization;
  * ADA treatment discontinuation;
In CD: The predictive value of an absolute and relative faecal calprotectin measured by IBDoc® between baseline and week 8 | 8 weeks
  The predictive value of an absolute and relative faecal calprotectin measured by IBDoc® between baseline and week 8 in predicting:
  * steroid-free clinical remission at week 26, without prior need for ADA dose optimization;
  * steroid-free clinical response (HBI <5 or drop in HBI with ≥3) at week 12, and week 26, without prior need for ADA dose optimization;
  * steroid-free biological remission (CRP <5 mg/L) at week 12, and week 26, without prior need for ADA dose optimization;
  * steroid-free biological response (CRP <5 mg/L or drop with ≥50%) at week 12, and week 26, without prior need for ADA dose optimization;
  * ADA treatment optimization;
  * ADA treatment discontinuation;
In UC and CD: correlations with IBDoc® measurements of faecal calprotectin and ELISA measurements of faecal calprotectin, different components of the Mayo score, C reactive protein and serum albumin | 26 weeks
  The correlation between IBDoc® measurements of faecal calprotectin, ELISA measurements of faecal calprotectin, different components of the Mayo score, C reactive protein and serum albumin, at weeks 0, 4, 8, 12 and 26;
In UC and CD: The convenience of the IBDoc® system to the patient and the health care professional | 26 weeks
  The convenience of the IBDoc® system for patients, and health care professionals

CONTACTS AND LOCATIONS:
Overall Officials: Marc Ferrante, MD PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- UZ Leuven, Leuven, Belgium